CLINICAL TRIAL: NCT03472729
Title: AGE-ON 2.0: Expanding and Evaluating a Tablet Training Program for Older Adults
Acronym: AGEON2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 3670
Record Dates: First submitted 2017-09-19; First posted 2018-03-21 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2019-08

CONDITIONS: Social Isolation
Keywords: Social isolation; Older adults; Technology
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AGE-ON Workshop (Experimental): Intervention participants will take part in a 6-week workshop to learn 1) basic features of the iPad; 2) how to use the internet; 3) how to take and view photos; 4) how to send and receive emails; and 5) other 'fun' functions.
  Interventions: Other: AGE-ON Workshop
- Wait-list control (No Intervention): Wait-list control group to be offered workshops after the study is complete

INTERVENTIONS:
Other: AGE-ON Workshop — Series of workshops to reduce social isolation through technology use.
  Arms: AGE-ON Workshop

SUMMARY:
AGE-ON is a series of workshops developed by the Regional Geriatric Program central, based in Hamilton, Ontario. The goal of these workshops is to teach older adults with limited computer knowledge how to use tablet computers to connect with friends and family and gather information related to issues of importance to them. The overwhelming positive response to three initial pilots proved the interest in such a program from seniors in the community. Preliminary feedback from program participants was collected as part of the initial pilot; the investigators would now like to use this feedback to improve the existing workshops and expand implementation of the program to a diverse population of older adults. The objective of this study is to conduct a formal mixed-methods evaluation of the updated AGE-ON workshops implemented at multiple community-based sites.

DETAILED DESCRIPTION:
Adults over 65 years are the fastest growing segment of Canada's population. Social isolation (defined as living alone with infrequent social contact and/or few social network ties) and loneliness (a dissatisfaction with the discrepancy between desired and actual social connections) are of growing concern, as individuals are living longer and often living alone or far from family and close friends. Both loneliness and social isolation are related to poor quality of life and overall well being. The internet and communication technology may be important tools to help older adults connect with family and friends, thus maintaining or even enhancing social connections. They help users overcome physical and spatial barriers to connect with others. However many older adults have obstacles to internet and technology use such as lack of knowledge and efficacy, and concerns over privacy.

AGE-ON is a series of volunteer-run workshops developed in 2014 by the Regional Geriatric Program in Hamilton. The goal of these workshops is to teach older adults with limited computer knowledge how to use tablet computers to connect with friends and family and gather information related to issues of importance to them. Over six weeks, participants learn 1) basic features of the iPad; 2) how to use the internet; 3) how to take and view photos; 4) how to send and receive emails; and 5) other 'fun' functions. An initial pilot project conducted in 2014-2015 displayed an overwhelmingly positive response to the AGE-ON workshops by both participants and volunteers, generating local media attention and resulting in a large number of interested older adults being placed on a wait-list for future workshops. This response proved the interest and need for a program of this type in the community. Preliminary feedback was gathered from participants; the investigators would now like to use this feedback to improve and expand upon the existing curriculum, and conduct a formal evaluation of the workshops.

Through this randomized controlled trial the study team will conduct a formal evaluation of the AGE-ON workshops. Tablet and internet use and self-efficacy, barriers to technology use, social isolation, loneliness and quality of life will be assessed before and after the workshops. Qualitative feedback from participants will be collected after each workshop, and in-person and telephone interviews will be conducted with participants at the end of the workshops.

Based on preliminary findings from AGE-ON Level 1 pilot project, we expect that participants in the AGE-ON program will improve self-efficacy in using their tablet for variety of tasks, specifically communicating with family and friends, and accessing health information. We anticipate this will result in a reduction in social isolation and loneliness, and improvement in quality of life. We also expect that this benefit will extend beyond the individual participant themselves, to family members and friends of workshop participants. At the community-level, this project will establish partnerships between researchers at McMaster University (Portal team), clinicians (Regional Geriatric Program, central) and organizations that work with older adults in the community (YWCA, assisted living facilities).

ELIGIBILITY:
Inclusion Criteria:

* Interest in participating in a tablet training workshop
* Read, speak and understand English

Exclusion Criteria:

* Previous participation in AGE-ON pilot

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Duke Social Support Index | 6-weeks
  To understand the impact of AGE-ON on participants' social isolation

SECONDARY OUTCOMES:
de Jon Gierveld Loneliness Scale | 6 weeks
  To understand the impact of AGE-ON on participants' loneliness
CASP-12 | 6 weeks
  Quality of life

OTHER OUTCOMES:
Participant satisfaction | 6 weeks
  Collected from participant feedback on a Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Neil-Sztramko, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neil-Sztramko SE, Coletta G, Dobbins M, Marr S. Impact of the AGE-ON Tablet Training Program on Social Isolation, Loneliness, and Attitudes Toward Technology in Older Adults: Single-Group Pre-Post Study. JMIR Aging. 2020 Apr 20;3(1):e18398. doi: 10.2196/18398. PMID 32310146